CLINICAL TRIAL: NCT00081822
Title: A Phase I Study of Clofarabine & Cytosine Arabinoside Therapy for Older Adults With Acute Myeloid Leukemia
Brief Title: Study of Clofarabine & Cytosine Arabinoside Therapy for Older Adults With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F040114019; UAB 0341 (Other: Institutional study protocol number)
Record Dates: First submitted 2004-04-21; First posted 2004-04-23 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Foran; clofarabine; cytosine arabinoside; acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine + Ara-C (Other): An initial dose escalation of clofarabine with a fixed standard dose of Ara-C in phase I will be used to determine an optimal phase II dose.
  Interventions: Drug: clofarabine; Drug: Ara-C

INTERVENTIONS:
Drug: clofarabine — Clofarabine should be administered by daily intravenous infusion over 2 hours.Following demonstration of DLT at Dose Level -I (22.5 mg/m2/day days 2-6) and demonstration that Dose Level -II (15mg/m2day days 2-6) is the 'optimal phase II dose', an additional Dose Level -1½ (20mg/m2/day, days 2-6) will be added to explore an increased dose of clofarabine intermediate between Dose Levels -I and -II.
  Other Names: CLOFAREX TM
Drug: Ara-C — Ara-C: Administer Ara-C by continuous infusion of 100mg/m2/day on days 1 to 7 for cycle 1, and on days 1 to 5 for cycles 2 & 3.
  Other Names: Cytosine arabinoside; Cytarabine; Cytosar-U; Arabinosyl

SUMMARY:
The purpose of this study is to determine the recommended phase II dose of clofarabine when administered in combination with standard dose Ara-C to older (>=60 years of age) patients with newly diagnosed acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This phase I/II trial will include an initial dose escalation of clofarabine with a fixed standard dose of Ara-C in phase I to determine the 'optimal phase II dose'. Patients will be enrolled into phase I in cohorts of 3-6 beginning at Dose Level I of clofarabine (30 mg/m2/day, days 2-6). If 0/3 or 1/6 patients experience dose-limiting toxicity (DLT), clofarabine will be escalated to Dose Level II (40mg/m2/day, days 2-6). If >1/3 or ≥2/6 patients experience DLT on Dose Level II, then Dose Level I will be declared the optimal phase II dose. However, if 0/3 or 1/6 patients experience DLT on Dose Level II, then Dose Level II will be declared the optimal phase II dose. In the event that ≥2 patients experience DLT at Dose Level I, clofarabine will be dose reduced to Dose Level -I (22.5mg/m2/day, days 2-6). Accrual will continue in cohorts of 3-6 patients, in a phase I fashion. If 0/3 or 1/6 patients experience DLT, then Dose Level -I will be declared the 'optimal phase II dose'. In the event that ≥2 patients experience DLT at Dose Level -I, clofarabine will be further dose reduced to Dose Level -II (15mg/m2/day, days 2-6). Accrual will again proceed in cohorts of 3-6 patients. If 0/3 or 1/6 experience DLT, then Dose Level -II will be declared the 'optimal phase II dose'. In the event that ≥2 patients experience DLT at Dose Level -II, accrual to the protocol will be halted.

Enrollment will proceed at the optimal phase II dose in a Simon 2-stage design to determine the CR rate and treatment-related mortality initially in 16 patients; if the CR rate and TRM is acceptable , then enrollment will continue to approximately 46 patients or until complete.

Induction Therapy (cycle 1)

* 7 day cycle Day 1 Aggressive Hydration x12-24hrs, followed by Ara-C 100mg/m2/day by 24hr IV continuous infusion days 1-7
* PK analysis Ara-C alone on Day 1 (plasma & intracellular) Day 2 Dexamethasone 10mg IV QD prior to clofarabine days 2-6 Clofarabine 2 hour daily infusion days 2-6
* PK analysis of Ara-C & clofarabine on Day 2
* Bone Marrow Apoptosis analysis (plasma & intracellular) Day 3 *Bone Marrow Apoptosis analysis (plasma & intracellular) Day 6 *PK analysis of Ara-C and clofarabine (plasma only) (UAB only) Day 8 Initiation of prophylactic antibiotic, antifungal & antiviral therapy Day 15 *QOL analysis Day 15-22 Restaging BM Re-Induction if appropriate (see below) Day 16 GM-CSF 250μg/m2 daily until ANC >1,500/μl (if D15 BM aplasia, no residual AML) Day 28-49 Outcome BM, assessment of response Re-Induction (PR) or Post-Remission therapy (CR)
* QOL analysis 2 weeks after hospital discharge (approximately Day 42)

Re-Induction (cycle 2 if appropriate) (if Partial Remission after Induction, day 15-49) *5 day cycle Aggressive Hydration x12-24hrs Day 1 Dexamethasone 10mg IV QD days 1-5 Day 1 Clofarabine 2 hour daily infusion days 1-5 Day 1 Ara-C 100mg/m2/day days 1-5 (begin 4 hours after end of clofarabine infusion) Day 7 GM-CSF 250μg/m2 daily may be used until recovery ANC >1,500/μl Day 7 Initiation of prophylactic antibiotic, antifungal & antiviral therapy

Post-Remission Therapy (cycles 2 & 3 if appropriate) (if Complete Remission after Induction; must have ANC>1,000/μl , platelets >100/μl)

*5 day cycle Aggressive Hydration x12-24hrs Day 1 Dexamethasone 10mg IV QD days 1-5 Day 1 Clofarabine 2 hour daily infusion days 1-5 Day 1 Ara-C 100mg/m2/day days 1-5 (begin 4 hours after end of clofarabine infusion) Day 7 GM-CSF 250μg/m2 daily may be used until recovery ANC >1,500/μl Day 7 Initiation of prophylactic antibiotic, antifungal & antiviral therapy

Follow-up Monthly x 12 months 3-monthly x 2 years 4-monthly x 1 year 6-monthly x 1 year Annually thereafter

ELIGIBILITY:
Inclusion Criteria:

* Have newly diagnosed AML (FAB classification types M0-M2 or M4-M7 or WHO classification) excluding acute promyelocytic leukemia (APL) or AML with any of the following chromosomal translocations: t(15;17)(q22;q21); t(11;17)(q23;q21); t(11;17)(q13;q21); t(5;17)(q32;q12)..
* Have greater than or equal to 20% blasts in the bone marrow.
* Have greater than or equal to 20% cellularity in the bone marrow.
* Provide written informed consent.
* Must be 60-75 years of age at diagnosis.
* Have an Karnofsky performance status of ≥60.
* Women of childbearing potential (<1 year post-menopausal unless surgically sterilized) and sexually active males must have a negative urine pregnancy test, and agree to use an effective barrier method of birth control (i.e. latex condom, diaphragm, cervical cap, etc) to avoid pregnancy.
* Able to comply with study procedures and follow-up examinations.
* Have adequate organ function as indicated by the following laboratory values, obtained within 7 days prior to registration:

Parameter Required Value (IS units) Renal Serum creatinine <1.1 mg/dL Hepatic Serum bilirubin <2 x ULN AST and ALT ≤5 x ULN ULN = Institutional Upper Limit of Normal. Inclusion Laboratory Values

Exclusion Criteria:

* Patients with pre-existing myelodysplastic syndrome, or with antecedent hematologic disorder of >3 months duration, will be excluded. Those with concomitant myelodysplasia/trilineage dysplasia noted at the time of diagnosis of AML will be eligible 74
* Have secondary AML (AML following chemotherapy or radiation therapy).
* Have an active, uncontrolled systemic infection considered opportunistic, life threatening, or clinically significant at the time of treatment.
* Have a psychiatric disorder(s) that would interfere with consent, study participation or follow-up.
* Are receiving other chemotherapy or corticosteroids (unless the latter is administered at a low dose for pre-medication purposes or for the treatment of chronic conditions - e.g., rheumatoid arthritis).
* Have received prior treatment for leukemia. Patients who have received growth factors, cytokine support, leukapheresis, hydroxyurea, or cranial irradiation will be allowed but must discontinue treatment at least 24 hours prior to beginning treatment with clofarabine. If used, hydroxyurea must be discontinued 48 hours prior to the initiation of chemotherapy.
* Have any other severe concurrent disease (severe coronary artery disease (NYHA class >II), significant neurological disorder, uncontrolled diabetes, etc.), which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Have active central nervous system involvement with leukemia.
* Other malignancy within the past year, with the exception of basal cell or non-metastatic squamous cell carcinoma of the skin

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-01; Primary Completion 2009-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Median time to complete response (CR) | 1 year

SECONDARY OUTCOMES:
To evaluate quality of life parameters before, during and after therapy in the older adult (>60 years) population | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James M Foran, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The University of Nebraska, Omaha, Nebraska
  - The Cleveland Clinic Foundation, Cleveland, Ohio